CLINICAL TRIAL: NCT04727034
Title: A Multicenter, Randomized, Single-blind, Parallel Controlled Clinical Study on the Efficacy and Safety of Remimazolam Tosylate for Sedation in Gastroscopy
Brief Title: Efficacy and Safety of Remimazolam Tosylate for Sedation in Gastroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai East Hospital (Other); Affiliated Hospital of Jiaxing University (Other); The Second Affifiliated Hospital of Jiaxing University (Unknown); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, diansan su, Vice Chair of the Department of Anesthesiology, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: sudiansan1215
Record Dates: First submitted 2021-01-14; First posted 2021-01-27 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Hypoxia; Gastric Cancer; Sedation Complication; Propofol Adverse Reaction
Keywords: Hypoxia; Efficacy and Safety; Gastroscope; Remimazolam; Propofol
MeSH Terms: conditions — Hypoxia; Stomach Neoplasms | interventions — 4-methylbenzenesulfonic acid; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Propofol（1.5mg/kg）
  Interventions: Drug: Propofol
- Test group 1（Remimazolam tosylate 0.15mg/kg） (Experimental): Remimazolam tosylate 0.15mg/kg
  Interventions: Drug: Remimazolam tosylate
- Test group 2（Remimazolam tosylate 0.2mg/kg） (Experimental): Remimazolam tosylate 0.2mg/kg
  Interventions: Drug: Remimazolam tosylate

INTERVENTIONS:
Drug: Remimazolam tosylate — Remazolam tosylate is an ultra-short-acting benzodiazepine drug, which has a mild inhibitory effect on the respiratory and circulatory systems and has anterograde amnesia. These advantages make remazolam tosylate very likely to replace propofol in painless gastroscopic anesthesia.
  Arms: Test group 1（Remimazolam tosylate 0.15mg/kg）; Test group 2（Remimazolam tosylate 0.2mg/kg）
Drug: Propofol — Propofol is the most commonly used intravenous anesthetic for painless gastroscopy, but propofol significantly inhibits the respiratory and circulatory systems. Therefore, the incidence of intraoperative hypoxemia and hypotension is high.
  Arms: Control group

SUMMARY:
Propofol is the most commonly used intravenous anesthetic for painless gastroscopy, but propofol significantly inhibits the respiratory and circulatory systems. Therefore, the incidence of intraoperative hypoxemia and hypotension is high. Remazolam tosylate is an ultra-short-acting benzodiazepine drug, which has a mild inhibitory effect on the respiratory and circulatory systems and has anterograde amnesia. These advantages make remazolam tosylate very likely to replace propofol in painless gastroscopic anesthesia.

ELIGIBILITY:
Inclusion Criteria:

- 1)18≤age≤60 years old, no gender limit; 2) Patients receiving routine gastroscopy diagnosis and treatment; 3) ASA score is I or II; 4) 18 kg/m2<BMI<28kg/m2； 5) It is estimated that the operation time of gastroscope will not exceed 30 minutes; 6) Clearly understand, voluntarily participate in the research, and be signed and informed consent.

Exclusion Criteria:

1. Need to perform complicated endoscopic diagnosis and treatment techniques (such as cholangiopancreatography Surgery, endoscopic ultrasonography, endoscopic mucosal resection, endoscopic submucosa Stripping, oral endoscopic muscle dissection, etc.);
2. Patients who intend to undergo tracheal intubation;
3. It is judged to be difficult to manage the respiratory tract (modified Mallampati score is IV)patient;
4. Anemia or thrombocytopenia,( Hb<90g/L, PLT<80×109/L);
5. Diagnosed lung diseases (asthma, bronchitis, COPD, Pulmonary bullae,pulmonary embolism, pulmonary edema, lung cancer);
6. Liver and kidney disease;( AST and/or ALT≥2.5×ULN,TBIL≥1.5×ULN, blood creatinine is greater than the upper limit of normal);
7. There is a history of drug and/or alcohol abuse within 2 years before the beginning of the screening period.The average daily alcohol consumption exceeds 2 units of alcohol (1 unit = 360 mL beer Liquor or 45 mL liquor with 40% alcohol content or 150 mL grapes liqueur);
8. Hypertensive patients whose blood pressure has not been satisfactorily controlled by antihypertensive drugs(Sitting systolic blood pressure ≥160 mmHg during screening period, and/or diastolic pressure during screening period Pressure ≥100 mmHg);
9. Sitting systolic blood pressure ≤90 mmHg during the screening period;
10. Women who are pregnant or breastfeeding;
11. Benzodiazepines, opioids, propofol, lidoca Those who are allergic or contraindicated due to their drug components;
12. Participated in other drug clinical trials as subjects in the past 3 months;
13. The investigator believes that it is not appropriate to participate in this trial;
14. A well-diagnosed heart disease (heart failure, angina pectoris, myocardial infarction, heart rhythmabnormalities etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1800 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
The success rate of remazolam tosylate for sedation in gastroscopy diagnosis and treatment | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  1) Complete the entire process of gastroscopy; 2) No sedative remedy is given; 3) After the initial dose of the test drug is administered, additional administration ≤ 2 times within any 5-minute period; 4) The initial dose of propofol After the end, within any 5-minute period of additional administration ≤ 2 times, it is recorded as propofol (control group) successfully sedated

SECONDARY OUTCOMES:
Sedation induction time | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  induction time
Sedation recovery time | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  recovery time
Incidence of drug injection pain | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  drug injection pain
Doctor satisfaction and patient satisfaction | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  There is a scale from 1 to 10. Endoscopists and patients will score their satisfaction with the scale ,with 1-3 (dissatisfied),4-6 (satisfied) and 7-10 (very satisfied) after gastroscopy.
The time it takes for the patient to wake up and leave the hospital if the Sedation/Anaesthesia Discharge Rating Scale score exceeds 9 points; | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Sedation/Anaesthesia Discharge Rating Scale
The incidence of hypoxia during sedation | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  (75% ≤ SpO2 < 90% for <60 s)；(SpO2 < 75% for any duration or 75% < SpO2 < 90% for >/=60 s)
Other adverse events assessed by the World SIVA adverse sedation event reporting tool | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force and HFNC supportive oxygen therapy-related adverse events.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Renji Hospital, Shanghai, Shanghai, China
  - Shanghai East Hospital, Shanghai, Shanghai, China
  - Affiliated Hospital of Jiaxing University, Jiaxing
  - The Second Affifiliated Hospital of Jiaxing University, Jiaxing
  - The First Affiliated Hospital of Nanchang University, Nanchang

REFERENCES:
- [Derived] Zhu H, Su Z, Huai X, Chen C, Zhang X, Zhou J, Su D. Efficacy and safety of remimazolam tosylate for sedation during upper gastrointestinal endoscopy: study protocol for a multicenter randomized controlled trial. Trials. 2022 Dec 12;23(1):995. doi: 10.1186/s13063-022-06935-0. PMID 36510290